CLINICAL TRIAL: NCT02601352
Title: Characterization and Health Risk Assessment of Exposure to Source-Specific PM2.5 in Subjects in Beijing
Brief Title: Air Pollution and Cardiometabolic Study
Status: Completed | Type: Observational
Sponsor: WeiHuang (Other)
Responsible Party: Sponsor-Investigator, WeiHuang, Principal Investigator, Peking University
Organization: Peking University (Other)
Other Study IDs: WHuang15_17
Record Dates: First submitted 2015-11-03; First posted 2015-11-10 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Cardiovascular Outcomes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood and urine
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The study mainly focuse on examining the subjects living in traffic polluted area and assessing the popuation health risk using disease and risk assessment models.

ELIGIBILITY:
Inclusion Criteria:

* Living in PU community neighborhood，Non smoker and No diseases ,and so on.

Exclusion Criteria:

* Advanced microvascular or neuropathic complications and active cardiovascular disease,and so on.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Living in PU community neighborhood,Beijing, China
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2015-09; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Vascular endothelial function | Four months
  Vascular endothelial function measured by Endo-PAT2000
Arrythmias | Four months
  Twenty four-hour electrocardiograms

SECONDARY OUTCOMES:
System inflammatory | Four months
  Analyzed systemic inflammation biomarkers,such as C-reaction Protein and Blood coagulation by ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Wei Huang, PhD, Principal Investigator — Peking University School of Public Health
Locations (2):
- China (2):
  - Peking University ,School of Public Health, Beijing, Beijing Municipality
  - Peking University, Beijing, Beijing Municipality